CLINICAL TRIAL: NCT03163511
Title: An Open-Label, First-In-Human Study Evaluating the Safety, Tolerability, and Efficacy of VC-02™ Combination Product in Subjects With Type 1 Diabetes Mellitus and Hypoglycemia Unawareness
Brief Title: A Safety, Tolerability, and Efficacy Study of VC-02™ Combination Product in Subjects With Type 1 Diabetes Mellitus and Hypoglycemia Unawareness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ViaCyte (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); Horizon 2020 - European Commission (Other); Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: VC02-101
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia

STUDY DESIGN:
Intervention Model Description: There are two Cohorts in this study design. Cohort 1 was to enroll up to 15 subjects total. After Cohort 1 enrollment was completed, Cohort 2 was to enroll up to an additional 60 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): VC-02 Combination Product:
  Up to ten (10) VC-02-20 implants and up to two (2) VC-02-300 implants
  Interventions: Combination Product: VC-02 Combination Product
- Cohort 2 (Experimental): VC-02 Combination Product; Up to twelve units implanted of which up to ten (10) are VC-02-300 implants and the rest are VC-02-20 implants.
  Interventions: Combination Product: VC-02 Combination Product

INTERVENTIONS:
Combination Product: VC-02 Combination Product — PEC-01 cells loaded into a Delivery Device
  Other Names: PEC-Direct

SUMMARY:
VC02-101 will evaluate an experimental cell replacement therapy intended to provide a functional cure to subjects with Type 1 Diabetes and Hypoglycemia Unawareness.

DETAILED DESCRIPTION:
The purpose of this trial is to test if VC-02™ combination product can be implanted subcutaneously in subjects with Type 1 Diabetes and Hypoglycemia Unawareness and maintained safely for up to two years. It will also test if VC-02 is an effective treatment for these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women
* Diagnosis of T1DM for a minimum of five (5) years
* Hypoglycemia unawareness or significant glycemic lability
* Stable diabetic treatment
* Willingness to use a continuous glucose meter
* Acceptable candidate for implantation

Exclusion Criteria:

* History of islet cell, kidney, and/or pancreas transplant.
* Six (6) or more severe, unexplained hypoglycemic events within six (6) months of enrollment
* Uncontrolled or untreated thyroid disease or adrenal insufficiency
* Diabetic complications such as severe kidney disease or renal dysfunction, proliferative retinopathy, diabetic foot ulcers, amputations attributable to diabetes, and/or severe peripheral neuropathy
* Non-compliance with current anti-diabetic regimen
* Detectable stimulated serum C-peptide during screening period assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautham Marigowda, Study Director — Vice President, Clinical Development, Vertex
Locations (10):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - UCLA-UCI Alpha Stem Cell Clinic, Irvine, California
  - UC Davis - Alpha Stem Cell Clinic, Sacramento, California
  - University of California San Diego, San Diego, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio
- University Hospital Brussels, Brussels, Belgium
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keymeulen B, De Groot K, Jacobs-Tulleneers-Thevissen D, Thompson DM, Bellin MD, Kroon EJ, Daniels M, Wang R, Jaiman M, Kieffer TJ, Foyt HL, Pipeleers D. Encapsulated stem cell-derived beta cells exert glucose control in patients with type 1 diabetes. Nat Biotechnol. 2024 Oct;42(10):1507-1514. doi: 10.1038/s41587-023-02055-5. Epub 2023 Nov 27. PMID 38012450
- [Derived] Shapiro AMJ, Thompson D, Donner TW, Bellin MD, Hsueh W, Pettus J, Wilensky J, Daniels M, Wang RM, Brandon EP, Jaiman MS, Kroon EJ, D'Amour KA, Foyt HL. Insulin expression and C-peptide in type 1 diabetes subjects implanted with stem cell-derived pancreatic endoderm cells in an encapsulation device. Cell Rep Med. 2021 Dec 2;2(12):100466. doi: 10.1016/j.xcrm.2021.100466. eCollection 2021 Dec 21. PMID 35028608
- [Derived] Ramzy A, Thompson DM, Ward-Hartstonge KA, Ivison S, Cook L, Garcia RV, Loyal J, Kim PTW, Warnock GL, Levings MK, Kieffer TJ. Implanted pluripotent stem-cell-derived pancreatic endoderm cells secrete glucose-responsive C-peptide in patients with type 1 diabetes. Cell Stem Cell. 2021 Dec 2;28(12):2047-2061.e5. doi: 10.1016/j.stem.2021.10.003. PMID 34861146

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: VC-02 Combination Product:
  Up to ten (10) VC-02-20 implants and up to two (2) VC-02-300 implants
  VC-02 Combination Product: PEC-01 cells loaded into a Delivery Device
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 2 | 47
Completed | 1 | 14
Not Completed | 1 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 2 | 47 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 47 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (5.66) | 47.9 (9.19) | 47.2 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 22 | 23
  Male | 1 | 25 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 2 | 46 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 28 | 28
  Belgium | 0 | 5 | 5
  United States | 2 | 14 | 16
Duration of Type 1 Diabetes [Mean (Standard Deviation); unit: years] — Number of years from onset of type 1 diabetes to the informed consent date, rounded to the nearest integer.
  years | 20 (19.8) | 33.2 (13.65) | 32.7 (13.92)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All AEs in Cohort 1 Participants
Description: Incidence of all AEs and evaluation of causality related to VC-02 combination product, the surgical procedures, and the immunosuppressive drug regimen.
Time Frame: Enrollment (Visit 3, Day 1) through the Month 4 Visit
Measure: Number; unit: Adverse Events
Arm/Group | Cohort 1
Number analyzed (Participants) | 2
Adverse Events
  Total Adverse Events | 33
  Adverse Events Related to IP | 2
  Adverse Events Related to Surgical Procedure | 24
  Adverse Events Related to Immunosuppression | 8

2. Primary Outcome: Change in C-peptide for Cohort 2 Subjects
Description: Change from baseline to Week 26 in C-peptide area under the curve from 0 to 4 hours following a mixed meal tolerance test.
Time Frame: Baseline to Week 26 Visit
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Cohort 2
Number analyzed (Participants) | 42
ng*hour/mL | .1292 (.33157)

ADVERSE EVENTS:
Time Frame: Adverse events were reported for Cohort 1 participants from date of enrollment through week 26. Adverse events were reported for Cohort 2 participants from date of enrollment through week 104.
Description: AEs were reported on a CRF at visit 2 (Wk -4) and at every subsequent visit through end of study. The definitions used for classifying AEs/SAEs are consistent with clinicaltrials.gov definitions. Adverse Events of Special Interest (AESIs) are defined as AEs that lead to the unexpected or premature explantation of VC-02-300 or sentinel units, AEs that result in early withdrawal from study, and severe hypoglycemic events occurring after VC-02 implantation possibly or definitely related to VC-02.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/2 | 19/47
Other Adverse Events (participants affected / at risk) | 2/2 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=47)
Hematoma, post-procedural (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Diabetic Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse Drug Reaction (General disorders) | 0 (0) | 2 (2)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Norovirus (Infections and infestations) | 0 (0) | 1 (1)
Liver Abscess (Infections and infestations) | 0 (0) | 1 (1)
Parvovirus B19 Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision Site Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Operative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=47)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 14 (18)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (3)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 3 (4)
Vitreous floaters (Eye disorders) | 0 (0) | 2 (3)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (6)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 20 (33)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (4)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 19 (34)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 13 (18)
Adverse drug reaction (General disorders) | 0 (0) | 4 (6)
Application site discomfort (General disorders) | 0 (0) | 1 (1)
Application site rash (General disorders) | 0 (0) | 1 (1)
Application site vesicles (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 5 (6)
Chills (General disorders) | 0 (0) | 2 (3)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 14 (17)
Feeling jittery (General disorders) | 0 (0) | 1 (1)
Implant site extravasation (General disorders) | 0 (0) | 1 (4)
Implant site irritation (General disorders) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 0 (0) | 3 (3)
Infusion site bruising (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 7 (9)
Pain (General disorders) | 0 (0) | 3 (3)
Peripheral swelling (General disorders) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 5 (5)
Temperature intolerance (General disorders) | 0 (0) | 2 (2)
Vaccination site pain (General disorders) | 0 (0) | 3 (3)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 3 (3)
Sensitisation (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (2)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 3 (3)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 4 (4)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (4)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 12 (18)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Root canal infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 7 (13)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site discharge (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 6 (9)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (5) | 29 (53)
Incision site pruritus (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision site swelling (Injury, poisoning and procedural complications) | 0 (0) | 6 (7)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 11 (20)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 10 (11)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Post procedural pruritus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 6 (13)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 5 (8)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (2) | 6 (15)
Procedural pain (Injury, poisoning and procedural complications) | 1 (7) | 34 (110)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 8 (10)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 4 (6)
Blood magnesium decreased (Investigations) | 0 (0) | 2 (2)
Blood magnesium increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 2 (2)
Blood urea increased (Investigations) | 0 (0) | 1 (3)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Drug level above therapeutic (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2)
Immunosuppressant drug level increased (Investigations) | 0 (0) | 2 (2)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 6 (8)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — This non-serious, adverse event was classified as an Adverse Event of Special Interest (AESI). This hypoglycemic event was considered severe and possibly related to the IP.
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 16 (21)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (2)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 14 (18)
Device dislocation (Product Issues) | 0 (0) | 2 (2) — One (1) of the Device Dislocation, non-serious, adverse events was classified as an Adverse Event of Special Interest (AESI). The event was considered an AESI because it led to a premature explantation of a VC-02 unit.
Device extrusion (Product Issues) | 0 (0) | 3 (4) — Two (2) of the Device Extrusion, non-serious, adverse events were classified as Adverse Events of Special Interest (AESIs). The events were considered an AESIs because they led to premature explantation of VC-02 units.
Device power source issue (Product Issues) | 0 (0) | 1 (1)
Drug delivery system issue (Product Issues) | 0 (0) | 1 (1) — This event was classified as an AESI. One of the participant's implanted VC-02 units exhibited lumen expansion due to accumulation of cartilage, likely graft-derived. Device integrity was maintained. This event led to premature explantation.
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (5)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Poor quality sleep (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nipple exudate bloody (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (13)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fasciectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 4 (4)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT03163511/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT03163511/SAP_001.pdf